CLINICAL TRIAL: NCT05458245
Title: TIBOLA : Multicenter Descriptive Study in Eastern France
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elisabeth BAUX, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI121
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: TIBOLA; Rickettsia Infections
Keywords: dermacentor; DEBONEL
MeSH Terms: conditions — Spotted Fever Group Rickettsiosis; Rickettsia Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TIBOLA (TIck-BOrne LymphAdenopathy) is a tick-borne disease. The pathogen is most often rickettsia (R. slovaca or R. raoultii), but other strict intracellular bacteria have been described (Francisella tularensis, Coxiella burnetii, Bartonella hensenlae).

Transmitted by ticks (Dermacentor), it is characterized by an inoculation eschar at the tick bite site, accompanied by painful loco-regional lymphadenopathy. It is most often a benign pathology, which can nevertheless leave sequellar alopecia or persistent asthenia.

In spring 2021, an impression of increased cases was reported by clinicians in Eastern France. The study aims to clarify the clinical-biological presentation and the evolution of the number of cases of TIBOLA in this region between 2016 and 2021.

At the same time, entomologists have noted an upsurge in this tick in certain biotopes in recent years.

ELIGIBILITY:
Inclusion Criteria:

* Person, minor or major,
* having been diagnosed with TIBOLA
* between January 1, 2016 and December 31, 2021
* at the University Hospital of Nancy or Strasbourg in the departments of infectious and tropical diseases, dermatology, microbiology and pediatrics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Definite case: clinically compatible (inoculation eschar with locoregional adenopathy(s) +/- general signs) +/- tick bite noted AND microbiological proof (positive PCR or seroconversion for a microorganism responsible for TIBOLA) OR
  * Probable case: clinically compatible (inoculation eschar with locoregional adenopathy(s) +/- general signs) AND tick bite noted without microbiological proof.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of cases of TIBOLA | baseline

SECONDARY OUTCOMES:
Epidemiological and demographic characteristics | baseline
  gender, age, habitat, hobbies, occupation
Characteristics of tick bites | baseline
  frequency, location, date
Frequency of the various symptoms and clinical signs of the disease | baseline
  inoculation ulcer, alopecia, lymphadenopathy, asthenia, fever, rash, headache, arthromyalgia, pruritus, facial oedema, other
Biological results | baseline
  serology and PCR of rickettsia, non-specific abnormalities
Treatment | baseline
  nature, efficiency
Entomological analysis | evolution between 2016 and 2021
  respective proportion of Dermacentor and Ixodes encountered on the territory. Detection by molecular biology of the presence of Rickettsia spp. in ticks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Yves Hansmann, Strasbourg
  - Elisabeth Baux, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Kotzyba J, Baux E, Hansmann Y, Boyer P, Jaulhac B, Martinot M, Martha B, Kaeuffer C, Bonijoly T, Bani-Sadr F, Legoff A, Hoefler F, Blot M, Bourdellon L, Zilliox L, Boulanger N, Lefevre B. Tick-borne lymphadenopathy in northeastern France: a human and vector clinical-epidemiological study. Parasit Vectors. 2025 Oct 24;18(1):428. doi: 10.1186/s13071-025-07078-2. PMID 41137175